CLINICAL TRIAL: NCT00786136
Title: Multicenter Randomized Controlled Study of Rosuvastatin for Prevention of Contrast Induced Acute Kidney Injury in Patients With Diabetes and Slight to Moderate Renal Insufficient
Brief Title: Rosuvastatin Prevent Contrast Induced Acute Kidney Injury in Patients With Diabetes
Acronym: TRACK-D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, MD, vice president, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SYNH-20081028
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Diabetes Mellitus; Chronic Kidney Disease
Keywords: diabetes mellitus; chronic kidney disease; contrast induced acute kidney injury; angiography
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency, Chronic | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): perioperative rosuvastatin administration for at least 5 dosages
  Interventions: Drug: rosuvastatin
- control (Placebo Comparator): blank control of perioperative statin administration
  Interventions: Drug: rosuvastatin

INTERVENTIONS:
Drug: rosuvastatin — rosuvastatin

SUMMARY:
The number of cardiac angiography and percutaneous coronary interventions (PCI) has increased steadily in recent years. This has resulted in the increasing incidence of contrast-induced acute kidney injury (CIAKI). Major risk factors for CIAKI include older age, diabetes mellitus (DM), chronic kidney disease(CKD), the concurrent use of nephrotoxic drugs, hemodynamic instability, etc. Importantly, DM appears to act as a risk multiplier, meaning that in a patient with CKD it amplifies the risk of CIAKI.

The aim of this multicenter prospective, randomized, controlled study is to evaluate whether statins treatment during the perioperative period would reduce the risk of CIAKI in a high-risk population of patients with both type 2 diabetes mellitus (T2DM) and CKD undergoing coronary angiography or noncoronary angiography, and evaluate the influence of such potential benefit on short-term outcome.

ELIGIBILITY:
Inclusion Criteria:

* Planned diagnostic coronary or peripheral artery angiography
* T2DM
* CKD stages 2 and 3, eGFR 30 to 89ml/min per 1.73m2
* Statin naive, or not on statin treatment for at least 14 days
* Withdrawal metformin or aminophylline for 48h before angiography
* Total iodixanol volume

Exclusion Criteria:

* Hypersensitivity to iodine-containing compounds and statins
* Type 1 diabetes mellitus
* Ketoacidosis
* Lactic acidosis
* CKD stages 1,4 or 5 (eGFR≥90ml/min per 1.73m2 or eGFR<30ml/min per 1.73m2)
* STEMI
* NYHA class IV or hemodynamic instability
* Administration of any iodinated CM within 14 days before randomization
* LDL-C<1.82mmol/L（70mg/dL）
* Hepatic dysfunction (ALT 3 times greater than upper normal limit)
* Thyreoid insufficiency
* renal artery Stenosis(unilateral >70％ or bilateral stenosis>50％)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2998 (Actual)
Dates: Start 2008-12; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
An absolute increase in SCr >=0.5mg/dL（>=44.2μmmol/L）or a >= 25% increase in SCr from baseline to 72h after the procedure | 72 h

SECONDARY OUTCOMES:
The composite of hospitalization for aggravated renal function, acute renal failure, dialysis or hemofiltration, aggravated at least 1 class of heart function, acute left ventricular failure or death from all causes. | 30 d

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD, Principal Investigator — Shenyang Northern Hospital
Locations (53):
- China (53):
  - The Armed Police General Hospital, Beijing, Beijing Municipality
  - The Chinese people's liberation army general hospital affiliated hospitals, Beijing, Beijing Municipality
  - Peking University first hospital, Beijing, Beijing Municipality
  - General Hospital Of The Second Artillery Force of the PLA, Beijing, Beijing Municipality
  - The General Hospital of the People's Liberation Army (PLAGH) ( Hospital 301), Beijing, Beijing Municipality
  - The Third Military Medical University, Chongqing Xinqiao Hospital, Chongqing, Chongqing Municipality
  - Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing, Chongqing Municipality
  - First Hospital of Lanzhou University, Lanzhou, Gansu
  - Dongguan Kanghua Hospital, Dongguan, Guangdong
  - General Hospital of Guangzhou Military Command of PLA, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong
  - Chinese People's Liberation Army 252th Hostipal, Baoding, Hebei
  - CanZhou Central Hospital, Cangzhou, Hebei
  - Shijiazhuang International Peace Hospital, Shijiazhuang, Hebei
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - HeNan Provincial People's Hospital, Zhengzhou, Henan
  - WuHan Asia Heart Hosital, Wuhan, Hubei
  - WuHan Union Hospital Of China, Wuhan, Hubei
  - TongJi Medical College HuaZhong University Of Science & Technology, Wuhan, Hubei
  - Renmin Hospital Of Wuhan University, Wuhan, Hubei
  - Wuhan General Hospital of Guangzhou Military Area Command of Chinese PLA, Wuhan, Hubei
  - Nanjing First Hospital, Nanjing, Jiangsu
  - NanJing Drum Tower Hospital, Nanjing, Jiangsu
  - FAW subsidiary of the General Hospital of Jilin University (Jilin University, Fourth Hospital), Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Changchun Central Hospital, Changchun, Jilin
  - General Hospital of Liaoning Anshan Iron and Steel Group Corporation, Anshan, Liaoning
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - Fushun central hospital, Fushun, Liaoning
  - The First Affiliated Hospital of Liaoning Medical College, Jinzhou, Liaoning
  - ShenZhou Hopital Of ShenYang Medical College, ShengYang, Liaoning
  - PLA 202 Hospital, Shenyang, Liaoning
  - Shenyang Nortern Hospital, Shenyang, Liaoning
  - Affiliated Hospital of LiaoNing University of Traditional Chinese Medicine, Shenyang, Liaoning
  - The Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - The 463th Hospital Of PLA, Shenyang, Liaoning
  - Affiliated Hospital of Ningxia Medical College, Yinchuan, Ningxia
  - General Hospital of Jinan Military Area Command of Chinese PLA, Jinan, Shandong
  - 88th Hospital of the Chinese PLA, TaiAn, Shandong
  - Ruijin Hospital Affiliated to the Medical College of Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Xijing Hospital of the Fourth Military Medical University, XiAn, Shanxi
  - Chengdu Military General Hospital, Chengdu, Sichuan
  - PLA 254 Hosipital, Tianjin, Tianjin Municipality
  - Affiliated Hospital Of Medical College Of The Chinese People's Armed Polic Forces, Tianjin, Tianjin Municipality
  - WuluMuqi General Hospital of PLA Lanzhou Military Area Command, Ürümqi, Xinjiang
  - The First Affilliated Hospital Of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kunming Medical College, Kunming, Yunnan
  - Kunming General Hospital of PLA, Kunming, Yunnan
  - The First Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang
  - Baotou city central hospital, Baotou
  - Baotou iron and steel group company worker hospital, Baotou

REFERENCES:
- [Derived] Li J, Li Y, Wang X, Yang S, Gao C, Zhang Z, Yang C, Jing Q, Wang S, Ma Y, Wang Z, Liang Y, Han Y. Age, estimated glomerular filtration rate and ejection fraction score predicts contrast-induced acute kidney injury in patients with diabetes and chronic kidney disease: insight from the TRACK-D study. Chin Med J (Engl). 2014;127(12):2332-6. PMID 24931252
- [Derived] Han Y, Zhu G, Han L, Hou F, Huang W, Liu H, Gan J, Jiang T, Li X, Wang W, Ding S, Jia S, Shen W, Wang D, Sun L, Qiu J, Wang X, Li Y, Deng J, Li J, Xu K, Xu B, Mehran R, Huo Y. Short-term rosuvastatin therapy for prevention of contrast-induced acute kidney injury in patients with diabetes and chronic kidney disease. J Am Coll Cardiol. 2014 Jan 7-14;63(1):62-70. doi: 10.1016/j.jacc.2013.09.017. Epub 2013 Sep 26. PMID 24076297